CLINICAL TRIAL: NCT04182893
Title: Clinical Study of ctDNA and Exosome Combined Detection to Identify Benign and Malignant Pulmonary Nodules
Acronym: ctDNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director,Endoscope Department,Shanghai Chest Hospital, Shanghai Chest Hospital
Other Study IDs: SHCHE201903
Record Dates: First submitted 2019-10-13; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Nodules
Keywords: bronchoalveolar lavage fluid; ctDNA; exosomes
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In this study, 12ml blood was extracted before bronchoscopy and 15ml bronchoalveolar lavage fluid was collected during bronchoscopy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary nodules population: We will enroll 300 pulmonary nodules penplein this study. After bronchoscopy, surgical examination or clinical follow-up, pulmonary nodules were finally diagnosed as malignant or benign.
  Interventions: Diagnostic Test: ctDNA and Exosome Combined Detection
- Healthy population: We will enroll 100 healthy penple in this study. After bronchoscopy, surgical examination or clinical follow-up, pulmonary nodules were finally diagnosed as malignant or benign.
  Interventions: Diagnostic Test: ctDNA and Exosome Combined Detection

INTERVENTIONS:
Diagnostic Test: ctDNA and Exosome Combined Detection — Through the detection and analysis of blood and alveolar lavage fluid of 300 patients with pulmonary nodules and 100 healthy population, the diagnostic efficacy of ctDNA and exosomes combined detceion will be studied.

SUMMARY:
This study through the detection of EGFR、ALK、ROS1、KRAS、HER2、BARF、NTRG1 seven ctDNA and exosome RNA in the blood and alveolar lavage of lung nodules patients and heavy smoking healthy population. If the results of ctDNA test is positive, the target nodule is malignant; if the reaults of ctDNA teste is negatie but exocome RNA is positive, the target nodule is also malignant. If the results of both tests are negtive, the target nodule is recognized as benign. The purpose is study the sensitivity, specificity and diagnostic accuracy of ctDNA and exosome combined detection in the identification of benign and malignant pulmonary nodules. Besides, the diagnostic efficacy of different specimens including blood and alveolar lavage in the identification of benign and malignant pulmonary nodules is also studied.

DETAILED DESCRIPTION:
Pulmonary nodules are round or irregular shape lesions with a diameter of less than or equal to 3cm. 10% lung nodules will become lung cancer, and lung cancer is evolved from small nodules.

Liquid biopsy is an effective and noninvasive means to assist in the early diagnosis of lung cancer, including circulating tumor cell、exosome and ctDNA detection. CtDNA is used to detect DNA fragments relesased to plasma by cracking or apoptotic tumor cells. Exosomes are derived from living cells, and researchers found that exosome nucleic acid detection of living cells may be closely related to the dynamic development of tumors.

This study through the detection of EGFR、ALK、ROS1、KRAS、HER2、BARF、NTRG1 seven ctDNA and exosome RNA in the blood and alveolar lavage of lung nodules patients and heavy smoking healthy population. If the results of ctDNA test is positive, the target nodule is malignant; if the reaults of ctDNA teste is negatie but exocome RNA is positive, the target nodule is also malignant. If the results of both tests are negtive, the target nodule is recognized as benign. The purpose is study the sensitivity, specificity and diagnostic accuracy of ctDNA and exosome combined detection in the identification of benign and malignant pulmonary nodules. Besides, the diagnostic efficacy of different specimens including blood and alveolar lavage in the identification of benign and malignant pulmonary nodules is also studied.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years old; The diameter of pulmonary lesions is 0.5-3cm in chest CT within 3 months; Healthy patients in normal control group had a smoking index ≥400; Patients who are eligible and intend to bronchoscopy.

Exclusion Criteria:

The patient received blood transfusion within 1 month； Patients suffer from autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, sjogren's syndrome, etc； Patients with cardiopulmonary dysfunction or other taboos, not suitable for bronchoscopy; Patients refused to participate in this clinical trial; The investigator considerates that the patient has other conditions that is unsuitable for this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study population include 2 groups: pulmonary nodules group and healthy people group.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficiency of ctDNA and exosome combined detection in the identification of benign and malignant pulmonary nodules. | 9 months
  Immunohistochemical method was used in ctDNA and exosome combined detection, to detect the blood and alveolar lavage of healthy people and patients with pulmonary nodules.Using the final diagnosis as the standard, the gene mutation threshold of benign and malignant lesions were demarcated, and the differences in gene expression between different types of diseases and the differences in diagnostic rates of blood and alveolar lavage fluid were explored.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided